CLINICAL TRIAL: NCT05133869
Title: BROCA-intervention Brain Outcome After Cardiac Arrest- Single Case Experimental Design Intervention Study
Brief Title: Brain Outcome After Cardiac Arrest - Intervention
Acronym: BROCA-i
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University (Other)
Collaborators: Rijnstate Hospital (Other); Adelante, Centre of Expertise in Rehabilitation and Audiology (Other); Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL77453.068.21
Record Dates: First submitted 2021-09-14; First posted 2021-11-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Heart Arrest, Out-Of-Hospital; Cognitive Impairment
Keywords: Cardiac Arrest; Cognitive Rehabilitation; Neuroplasticity; Cognitive training
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Cognitive Dysfunction; Heart Arrest

STUDY DESIGN:
Intervention Model Description: This is a randomized multiple baseline single case experimental design (SCED) intervention study.
Masking Description: All participants receive the same intervention, therefore there is no masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Baseline + intervention + follow up (Experimental): All participants receive the same treatment in the same order. First there is a phase without treatment, the baseline phase. The length of this phase is randomly assigned to each participant. Then all participants follow a 42 day intervention, in which direct training and metacognitive training is combined. Afterwards they have a follow-up period, this length of this period is counterbalanced with the length of the baseline period so that the full study adds up to 150 days.
  Interventions: Device: Metacognitive training + direct training

INTERVENTIONS:
Device: Metacognitive training + direct training — The intervention will consist of a combination of direct training of the impaired cognitive function(s) and metacognitive strategy training for 42 days (6 weeks). Direct training will be done with the computer program Rehacom for 20 minutes, 5 times a week. Metacognitive strategy training will be given on a weekly or biweekly basis (6-10 sessions) by a trained therapist at Adelante.
  Rehacom is a brain training program developed to improve a variety of cognitive functions with the use of game-like cognitive training modules. During the intervention the participant should train with Rehacom for approximately 600 minutes in total.
  In addition to the direct training, the participant receives six to ten sessions of metacognitive strategy training. During this training they are taught strategies by a therapist to improve their performance on the Rehacom modules and on daily life functioning. Each metacognitive strategy is linked to one of the Rehacom modules.
  Other Names: Rehacom

SUMMARY:
People who suffered a cardiac arrest are often have cognitive impairments. In this study the investigators test the effectiveness of an intervention, combining direct training and metacognitive training, in a single case experimental design (SCED).

DETAILED DESCRIPTION:
SUMMARY

Rationale: The survival rate of patients after cardiac arrest and resuscitation has increased considerably. A common consequence of cardiac arrest is ischemic-hypoxic brain damage leading to cognitive impairment. Currently, there is a lack of knowledge regarding effectiveness of treatments to improve outcomes of patients with cognitive impairment after a cardiac arrest.

Objective: The primary objective is to test effectiveness of cognitive rehabilitation therapy to improve functioning on problematic well-defined personalized behaviour that is caused by an objective cognitive impairments after OHCA. Secondary objectives are to test the generalisation of the effect of the intervention towards other aspects of daily living, to estimate the effect of the intervention on objective and subjective measures of cognitive functioning, participation in society, and quality of life, and to detect evidence of neuroplasticity in MRI data.

Study design: This is a randomized multiple baseline single case experimental design (SCED) intervention study.

Study population: The four to six participants included in this study will be patients surviving a cardiac arrest and cardiopulmonary resuscitation with remaining cognitive impairments at least 3 months after the cardiac arrest, who are motivated to adhere to the training program tested in this study.

Intervention: The intervention will consist of a combination of direct training of the impaired cognitive function(s) and metacognitive strategy training for 42 days (6 weeks). Direct training will be done with the computer program Rehacom to train the impaired cognitive domains, for 20 minutes 5 times a week. Metacognitive strategy training will be given on a weekly or biweekly basis (6-10 sessions) by a trained therapist as current care.

Main study parameters/endpoints: The primary outcome measure is the score on a Visual Analogue Scale (VAS) of the severity of the main, predefined daily life problem caused by objective cognitive impairment(s) that the participant is dealing with. The primary outcome measure will be collected by an App, through which the patient will receive questions on his / her telephone, daily. Answering will take less than one minute. Secondary outcome measures are daily obtained VAS scores on general and potential other daily life problems, and scores on neuropsychological tests and questionnaires that are obtained four times during the study, and MRI data obtained at two different time-points.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The investigators foresee no relevant additional risk of cognitive rehabilitation therapy and follow up in this study. Daily training and collection of outcomes will be challenging, but feasible, since the investigators will include motivated patients who will mostly judge the careful follow up as pleasant and attentive. MRI scanning is only performed in patients suitable for scanning, no contrasts are used. Potential benefit from participation in this study is follow up and treatment of cognitive impairments may lead to improved functional recovery after cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must be mentally competent and meet all of the following criteria:

* Objectified cardiac arrest between 3 months and 2 years before inclusion.
* Age 18 - 75
* Cognitive impairments objectified by a score on the Montreal Cognitive Assessment (MoCA) ≤ 26 or abnormal scores on a neuropsychological assessment caused by low scores (more than 1,5 standard deviation below the mean of the norm group) on memory, attention, and/or executive functioning tasks
* Living independently (with minor help)
* Experiencing difficulties with more complex daily tasks (e.g. doing groceries, following conversations, etc.)
* Motivated to improve cognitive functioning and to participate in the study
* Proficient in Dutch to understand instructions, follow the training program and fill in the questionnaires
* Patients with a treatment indication for cognitive rehabilitation (as decided by a psychiatrist)
* Written informed consent

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Neurodegenerative disorder, or another brain disease known to impact cognition, such as stroke or dementia
* Substance abuse impacting cognition
* Psychiatric disorder in need of treatment
* Uncorrected visual or auditory deficiencies
* Not in possession of a computer or lack of computer skills
* Severe amnesia or aphasia
* Illiteracy
* In case of MRI contra-indications, such as an ICD or metallic implants, patients will be excluded from the MRI sub-study. The full list of contraindications can be found in the article of Ghadimi and Sapra (2020).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2022-04-21 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Change in main daily problem | 85 measurements in 150 days
  A Visual Analogue Scale (VAS) from 0 to 100 with higher scores meaning a worse outcome, of the severity of the predefined daily life problem caused by an objective cognitive impairment that the participant is dealing with.

SECONDARY OUTCOMES:
Change in other daily problems | 85 measurements in 150 days
  This measure consists of a VAS from 0 to 100 with higher scores meaning a worse outcome, of other potential personal daily life problems caused by the objective cognitive impairment next to the primary outcome measure.
Change in general functioning | 85 measurements in 150 days
  This measure consists of a VAS from 0 to 100 with higher scores meaning a worse outcome, of the problems in general cognitive domains (memory, planning/complex tasks, and attention).

OTHER OUTCOMES:
Change in neuropsychological assessment score: Memory, Auditory Verbal Learning Test | < day 1 (before baseline), after baseline (day 15-35 depending on the randomisation), after intervention (day 57 - 77 depending on the randomisation), after follow-up (day 150)
  Before baseline (< day 1), immediately after baseline, after intervention, immediately after follow up. The patient has to remember a list of words. This measures immediate recall, retention, and recognition.
  Unit: amount of correct words recalled and recognized.
Change in neuropsychological assessment score: Memory, Rivermead Behavioural Memory Test-Stories | < day 1 (before baseline)
  Before baseline (< day 1). The patient has to try to remember a short newspaper article.
  Unit: amount of correct information given.
Change in neuropsychological assessment score: executive functioning, Digit Span backward | < day 1 (before baseline)
  Before baseline (< day 1): Digit Span backward (executive functioning).
  The patient has to repeat a row of numbers in the opposite order.
  Unit: length of the longest number sequence the patient completes successfully.
Change in neuropsychological assessment score: executive functioning, Letter Fluency task | < day 1 (before baseline), after baseline (day 15-35 depending on the randomisation), after intervention (day 57 - 77 depending on the randomisation), after follow-up (day 150)
  Before baseline (< day 1), immediately after baseline, immediately after intervention, immediately after follow-up.
  The patient is asked to name as many things as possible in 1 minute that start with a certain letter.
  Unit: amount of correct words named
Change in neuropsychological assessment score: attention, digit span forward | < day 1 (before baseline), after baseline (day 15-35 depending on the randomisation), after intervention (day 57 - 77 depending on the randomisation), after follow-up (day 150)
  Before baseline (< day 1), immediately after baseline, immediately after intervention, immediately after follow-up.
  The patient has to recall a sequence of number in the same order.
  Unit: length of the longest number sequence the patient completes successfully
Change in neuropsychological assessment score: attention, Digit Symbol coding task | < day 1 (before baseline)
  Before baseline (< day 1): Digit Symbol coding task (attention)
  The patient has to complete as many rows of symbols by giving them the corresponding digit within two minutes.
  Unit: The amount of symbols correctly coded within 2 minutes
Change in Questionnaires: cognitive complaints | < day 1 (before baseline), after baseline (day 15-35 depending on the randomisation), after intervention (day 57 - 77 depending on the randomisation), after follow-up (day 150)
  CLC_IC: Checklijst Cognitie-Intensive care questionnaire to assess cognitive complaints
  Range: 0 - 10, higher scores indicate a worse outcome.
Change in Questionnaires: memory complaints | < day 1 (before baseline), after baseline (day 15-35 depending on the randomisation), after intervention (day 57 - 77 depending on the randomisation), after follow-up (day 150)
  the Everyday Memory Questionnaire-revised (EMQ-r) for subjective memory complaints.
  Range: 0 - 52 , higher scores indicate a worse outcome
Change in Questionnaires: participation | < day 1 (before baseline), after baseline (day 15-35 depending on the randomisation), after intervention (day 57 - 77 depending on the randomisation), after follow-up (day 150)
  Utrecht Scale for Evaluation of Rehabilitation-Participation (USER-P)- restriction questionnaire measures participation.
  Range: 0 - 100, a higher score indicates better outcome
Change in Questionnaires: quality of life | < day 1 (before baseline), after baseline (day 15-35 depending on the randomisation), after intervention (day 57 - 77 depending on the randomisation), after follow-up (day 150)
  The Life Satisfaction Questionnaire (LiSat-9) measures quality of life.
  Range: 1-6, a higher score indicates better outcome
Change in MRI-data, DTI | before baseline (< day 1), after follow-up (day 150)
  These data will be used to assess brain structural and functional connectivity, including spatiotemporal characteristics of cerebral rearrangements that associate with cognitive recovery. During a ±30 minute scan, the investigators will collect measures of resting state functional connectivity and structural integrity of white matter tracts with blood oxygenation level-dependent (BOLD) MRI and diffusion tensor imaging (DTI) on a clinical 3T scanner. Functional connectivity will be expressed in a region-based way and at a whole network level. The architecture of neuronal fibers will be based on DTI-derived diffusion anisotropy, principle diffusion direction in white matter, and tractography algorithms.
Demographics; age | before baseline (< day 1)
  age in years
Demographics; level of education | before baseline (< day 1)
  level of education according to Verhage.
Demographics; handedness | before baseline (< day 1)
  handedness: left, right, or both
Demographics; Living situation | before baseline (< day 1)
  living situation: alone, with partner, with partner and children, with other residents.
Medical history; time since OHCA | before baseline (< day 1)
  the time since the OHCA in months
Medical history; ROSC | before baseline (< day 1)
  Time till return of spontaneous circulation in minutes
Medical history; cause OHCA | before baseline (< day 1)
  Cause of cardiac arrest
Medical history; hospitalization length | before baseline (< day 1)
  Duration of comatose state and hospitalization in days
Medical history; implantations | before baseline (< day 1)
  The presence of any implantations or objects in the body. If so, what kind of implantation/object?
Medical history; Comorbidity | before baseline (< day 1)
  Any other disorders or illnesses besides the OHCA.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline van Heugten, prof, Principal Investigator — Maastricht University
Locations (3):
- Netherlands (3):
  - Rijnstate Hospital, Arnhem, Gelderland
  - Adelante, Hoensbroek, Limburg
  - Maastricht University, Maastricht, Limburg

IPD SHARING:
Plan to Share IPD: No